CLINICAL TRIAL: NCT05314192
Title: Non-invasive Assessment of Inflammatory Markers MIP-1 Alpha and IL-6 in Saliva of Post Myocardial Infarction and Stage 4 Periodontitis Patients
Status: Completed | Type: Observational
Sponsor: Ajman University (Other)
Collaborators: A B Shetty Memorial Institute of Dental Science (Other)
Responsible Party: Principal Investigator, sudhir rama varma, Clinical Assistant Professor, Ajman University
Other Study IDs: ABSM/EC/29/2020
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Myocardial Infarction; Periodontal Diseases
Keywords: MIP-1 Alpha; IL-6; Myocardial infarction; Periodontal disease
MeSH Terms: conditions — Myocardial Infarction; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy: Healthy cohorts with no underlying systemic or periodontal disease
  Interventions: Diagnostic Test: salivary test
- stage 2 periodontitis: patients with periodontitis but no underlying systemic periodontal disease
  Interventions: Diagnostic Test: salivary test
- MI patients with stage 4 periodontitis: patients who had MI and having stage 4 periodontitis patients
  Interventions: Diagnostic Test: salivary test
- MI patients without periodontitis: patients who had MI without periodontitis
  Interventions: Diagnostic Test: salivary test

INTERVENTIONS:
Diagnostic Test: salivary test — saliva was assessed for MIP-1 alpha
Diagnostic Test: salivary test — saliva was assessed for IL-6

SUMMARY:
Periodontitis is an immunoinflammatory disease caused by microorganisms leading to sequential loss of the supporting structures of periodontium, resulting in periodontal pocket formation, gingival recession eventually leading to tooth loss.[1] A bacterial plaque is formed during the destructive changes of the periodontium which initiates a host of inflammatory and immune responses.[2] These inflammatory responses may also cause an increase in inflammatory activities in atherosclerotic lesions in the coronary arteries resulting in the increased risk of cardiovascular events like myocardial infarction.[3] Myocardial infarction (MI) is a cardiovascular condition that occurs when there is deprivation of oxygen in the heart muscle is due to the sudden interruption of the blood supply resulting from the coronary artery blockage by a plaque causing myocardial ischemia and cell death. Inflammation is pivotal in the initiation and progression of atherosclerosis. Various cytokines and chemokines are released during inflammation.[4] These inflammatory markers may have diagnostic potential for the detection of various inflammatory diseases.[5] Macrophages secrete macrophage inflammatory protein-1 alpha (MIP-1 alpha) which recruits inflammatory cells, inhibits stem cells, and activates bone resorption cells.[6] Interleukin-6 (IL-6) is produced in response to tissue injury and infection and contributes to the differentiation of B cells, the proliferation of T cells, and bone resorption.[7] The levels of these inflammatory markers are seen to be increased in inflammatory conditions, which include myocardial infarction and stage 4 periodontitis. Therefore, this study aims to assess the levels of these inflammatory markers in patients with myocardial infarction and periodontitis.

DETAILED DESCRIPTION:
This was a cross-sectional study involving the patients of the department of periodontics and department of cardiology.

Patients included in the study were categorized into four groups: (1) group 1-healthy subjects, (2) group 2-stage 4 periodontitis patients, (3) group 3- post-MI patients with stage 4 periodontitis, (4) group 4- post-MI patients without periodontitis.

The severity of the periodontitis was assessed by a periodontist. The diagnosis of acute MI was made by the cardiologists. Oral health assessment in acute MI patients was done at the subjects' bedside after stabilization of the patient, so as not to interfere with the ongoing medical treatment. Subjects' identification was kept confidential.

All samples were collected from patients admitted within 48 hours of their cardiac event. Patients were diagnosed as acute ST-elevation myocardial infarction (STEMI) based on the elevation of ST segments on the electrocardiogram(ECG) by 0.1mV in contiguous leads in patients with signs and symptoms of myocardial ischemia and/ or development of new left bundle branch block, along with increased cardiac biomarkers. Non-ST-elevation myocardial infarction (NSTEMI) was diagnosed in patients with signs and symptoms of myocardial ischemia and depression in ST-segment on the ECG or new Q wave pathology along with elevation of cardiac biomarkers.[8] Stage four periodontitis was diagnosed using the World Workshop 2017 classification.[9] Subjects who had undergone oral prophylaxis or periodontal surgery in the past 6 months were not included in the study. Smokers, pregnant women, lactating mothers, and those on medication (anti-microbial, non-steroidal anti-inflammatory drugs) in the past 3 months as well as those with other chronic systemic diseases were excluded from the study. These were all excluded as each would affect the levels of biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* subjects who had MI
* who had stage 4 periodontal disease

Exclusion Criteria:

* subjects who did not have MI
* subjects who had systemic disease other than MI
* subjects who had medication in the past 3 months
* smokers
* pregnant and lactating women

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients included in the study were categorized into four groups: (1) group 1-healthy subjects, (2) group 2-stage 4 periodontitis patients, (3) group 3- post-MI patients with stage 4 periodontitis, (4) group 4- post-MI patients without periodontitis.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
salivary test for MIP-1 alpha | 72 hours
  saliva was assessed for biomarker MIP-1 alpha among the 4 groups
salivary test for IL-6 | 72 hours
  saliva was assessed for biomarker IL-6 among the 4 groups

CONTACTS AND LOCATIONS:
Locations (1):
- AB shetty Institute of dental sciences, Mangalore, India

IPD SHARING:
Plan to Share IPD: Undecided
The link will be shared among researchers upon request